CLINICAL TRIAL: NCT03599323
Title: Prospective, Non-interventional, Post-marketing, Multi-center, Single-cohort, Safety (Questionnaire) Investigation of Empecid L Cream (Clotrimazole 1%)
Brief Title: Study on the Safety of the Approved Product Empedic L Cream During Its Routine Use (Active Ingredient is Clotrimazole 1%)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: SATO PHARMACEUTICAL , Ltd. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 19439
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Vaginal Candida
MeSH Terms: conditions — Candidiasis, Vulvovaginal | interventions — Clotrimazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Clotrimazole 1% (Empecid L Cream, BAYB5097): Patients who self-selected Empecid L Cream, and who will have pharmacist intervention prior to purchase.
  Interventions: Drug: Clotrimazole 1% (Empecid L Cream, BAYB5097)

INTERVENTIONS:
Drug: Clotrimazole 1% (Empecid L Cream, BAYB5097) — Consumers who self-select and are then deemed appropriate users of the product by the pharmacist for treatment of Vulvar itching with rash due to recurrent vaginal candida (only in patients previously diagnosed and treated by a doctor).

SUMMARY:
Researchers already did trials that showed Empecid L Cream worked for patients with Vaginal yeast infection who were in those trials. In this trial, they want to learn if consumers that use the cream under the guidance of a pharmacist have any medical problems during the trial

ELIGIBILITY:
Inclusion Criteria:

- Consumers who self-select and are then deemed appropriate users of the product by the pharmacist for treatment of Vulvar itching with rash due to recurrent vaginal candida (only in patients previously diagnosed and treated by a doctor).

Exclusion Criteria:

* Patient with first episode
* Patient with allergy to Empecid Cream (Clotrimazole)
* Patient under 15 years old/ beyond 60 years old
* Pregnant women or women who may possibly be pregnant
* Patient with diabetes
* Patient who repeats indicated symptom frequently, have recurrent episodes (once every month or two, or twice or more within 6 months).
* Patients who does not know whether it is a recurrence symptom
* Patients who have a fever, chills, lower abdominal pain, back or shoulder pain, colored or bloody vaginal discharge, fishy-smelling vaginal discharge, cessation of menses, irregular or abnormal bleeding from the vagina, or ulcer, edema or erosion in the vagina or vulva suggesting they may have a different disease.

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The primary population of interest is composed of subjects 15 years or older and under 60 years who purchase Empecid L Cream.
Sampling Method: Non-Probability Sample
Enrollment: 1033 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2021-07-07 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse event (AE) and serious adverse event (SAE) in consumers using Empecid L Cream. | Up to one month
Types of AE recorded in Questionnaire | Up to one month

SECONDARY OUTCOMES:
Patterns and way of use of Empecid L Cream recorded in Questionnaire | Up to one month

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the NCT number or Bayer Study ID in the search field — http://clinicaltrials.bayer.com/